CLINICAL TRIAL: NCT02088164
Title: Long-Term Outcome of Subjects With Elevated PSA in Healthy Taiwanese Men
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200809020
Record Dates: First submitted 2012-05-16; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: PSA,; asian men,; survival
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Healthy men: Healthy men who received PSA screening

SUMMARY:
To determine the long-term survival outcome of subjects who had various PSA levels at screening

ELIGIBILITY:
Inclusion Criteria:

* Health men who received PSA screening at NTUH and CGMH

Exclusion Criteria:

* Prior history of prostate cancer

Min Age: 41 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Taiwanese healthy men who are older than 40 years
Sampling Method: Non-Probability Sample
Enrollment: 27741 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Diagnosis of prostate cancer | 20 years (average)

SECONDARY OUTCOMES:
Cancer-specific death | 20 years (average)
Overall survival | 20 years (average)

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan